CLINICAL TRIAL: NCT00544024
Title: Mefloquine Bioequivalence Among Three Commercial Tablet Formulations in Peruvian Subjects With Uncomplicated Plasmodium Falciparum Malaria
Brief Title: Mefloquine Bioequivalence Among 3 Commercially Available Tablets.
Status: Completed | Type: Observational
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Naval Medical Research Center (U.S. Federal Agency); Universidad Peruana Cayetano Heredia (Other); Ministry of Health, Lima Peru (Unknown)
Other Study IDs: CDC-NCZVED-3620; DoD#31595
Record Dates: First submitted 2007-10-12; First posted 2007-10-16 (Estimated); Last update posted 2007-10-16 (Estimated); Status verified 2007-10

CONDITIONS: Malaria
Keywords: Mefloquine
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Whole blood was obtained for analysis, but has been subsequently disposed after completion of drug analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Reference: Lariam was administered as whole tablets with food and water at a dose of 25 mg/kg (15 mg/kg on the first day and 10mg/kg on the second day) along with artesunate at a dose of 4 mg/kg/day for three days under supervision by clinical staff
- T1: Mephaquin was administered as whole tablets with food and water at a dose of 25 mg/kg (15 mg/kg on the first day and 10mg/kg on the second day) along with artesunate at a dose of 4 mg/kg/day for three days under supervision by clinical staff
- T2: Mefloquine-AC Farma was administered as whole tablets with food and water at a dose of 25 mg/kg (15 mg/kg on the first day and 10mg/kg on the second day) along with artesunate at a dose of 4 mg/kg/day for three days under supervision by clinical staff

SUMMARY:
The objective of this study was to determine the bioequivalence among three commercial tablet formulations of MQ, i.e. Lariam, Mephaquin, and Mefloquine-(AC Farma) when given in combination with artesunate.

DETAILED DESCRIPTION:
Pharmacokinetic parameters were determined for mefloquine in whole blood from Peruvian subjects with uncomplicated falciparum malaria administered Mephaquin®, Mefloquine-AC Farma, and Lariam®. The Mefloquine-AC Farma arm comprised 13 patients while the reference (Lariam) and Mephaquin arms consisted of 12 patients. Although Cmax was significantly less (p=0.04) in the Mephaquin arm (AUC0-t = 2500 ng/ml/day) relative to the reference (AUC0-t = 2820 ng/ml/day) arm, there were no significant differences in the AUC∞, tmax, and t1/2 for Mefloquine-AC Farma or Mephaquin relative to the reference. Except for the Cmax of the Mefloquine-AC Farma, the 90% confidence intervals for all parameters of both treatments were outside the specified FDA range of 80-125%. Therefore both formulations were not considered bioequivalent to the reference.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for enrolling patients included; male or non-pregnant female ≥ 18 years of age, infection with P. falciparum alone, with a parasite density between 250 and 50,000 asexual parasites/mm3 as determined by microscopic examination of a thick blood smear, informed consent from patient, and a willingness to be hospitalized for the first 24 hours after therapy is initiated and to return for follow-up visits through day 56.

Exclusion Criteria:

* Patients exhibiting evidence of severe malaria or with a history of an underlying chronic disease or illness that could interfere with the absorption of MQ, a history of hypersensitivity to MQ, or a history of neuropsychiatric illness or cardiac conduction problems were excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Thirty-nine adult subjects were initially enrolled in the study ranging in age from 18-61 years with a mean of 36 years. Seventy-two percent of the volunteer patients were male.
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2004-03; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Measure concentrations of mefloquine in blood to determine pharmacokinetic parameters and assess bioequivalence. | 56 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Green, PhD, Principal Investigator — Centers for Disease Control and Prevention; Wilmer Marquino, MD, Principal Investigator — Instituto Nacional de Salud, Lima, Peru; David Bacon, PhD, Principal Investigator — Naval Medical Research Center Detachment
Locations (1):
- Apoyo Hospital, Iquitos, Peru